CLINICAL TRIAL: NCT04959045
Title: The Effect of Flipped Classroom Teaching Method on the Academic Achievement and Skill Learning Level of Nursing Students in Skills Education
Brief Title: The Effect of Flipped Classroom Teaching Method on Academic Achievement and Skill Learning Level in Skills Education
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Nesrin Ogurlu, Lecturer- PhD Student, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Skills Training in Nursing
Record Dates: First submitted 2021-06-27; First posted 2021-07-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Nursing Students; Education
Keywords: Skills Training; Flipped Classroom Teaching; Academic Success

STUDY DESIGN:
Intervention Model Description: This research is a randomized controlled experimental study. It was planned to divide the students into two groups as experimental and control groups. Simple random sampling method will be used to determine the experimental and control groups. To ensure randomization, each student will be numbered and data sets (experiment and control) will be created.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Flipped Teaching Method Group) (Experimental): Intervention group students will be given skill training with the Flipped Teaching method.
  Interventions: Other: intervention group (Flipped Teaching Method Group)
- Control group (Traditional Method Group) (No Intervention): Control group students will receive skill training with the traditional method. No intervention will be made.

INTERVENTIONS:
Other: intervention group (Flipped Teaching Method Group) — Students will be given skill training with the Flipped Teaching method, which consists of outside and in-class applications.
  Out-of-Class Practice: A Learning Management System-Web-Based Distance Education System will be created for the Flipped Teaching method. Theoretical course topics and skill training videos will be uploaded to the system 7 days before the course day. Students will be able to watch the video tutorials in the number and frequency they want until the day of the lesson. At the end of the lesson, the mini-exam will be uploaded to the system.
  In-class practice: The researcher will come to the lesson prepared for classroom activities such as "question and answer". Theoretical lectures and skill demonstrations will not be made by the researcher. The researcher will only guide the students. Then, the students will be provided to perform the skill under the guidance of the researcher in the clinical skills laboratory.
  Arms: intervention group (Flipped Teaching Method Group)

SUMMARY:
In this study, it was aimed to determine the effect of the Flipped Classroom Teaching Method on the academic achievement and skill learning levels of nursing students in nursing skills education.

DETAILED DESCRIPTION:
Due to the rapid changes in science and technology, the increase in the number of students in higher education and the decrease in resources, the fact that students are in the Y and Z generation, who know the use of technology well, have advanced thinking and a rapid knowledge acquisition process, they are different from traditional teaching methods due to the Covid 19 pandemic. The use of teaching methods has become more important. In nursing education, the curriculum should support high-level learning, encourage active learning, education should be student-centered, and students should take responsibility for learning.

The traditional classroom model learning approaches, in which the student is a passive participant and under the control of the teacher, have been changing recently with the effect of new educational technologies, learner characteristics and learning expectations, and methods in which students are more active are needed. This change reveals structuring in the direction of the use of out-of-class time. One of these embodiments is the flipped classroom model. Presenting in-class activities to students outside the classroom in flipped classrooms is defined as bringing homework and activities that are expected to be done outside the classroom in the traditional structure. In the flipped learning model, the student reaches the basic level of knowledge outside the classroom, and spends the classroom time with high-level skills such as discussion, practice and problem solving.

In this study, it was aimed to determine the effect of the Flipped Classroom Teaching Method on the success of the students and the level of skill learning in skill education, which has an important place in nursing education. With the Flipped learning method, it is aimed to raise individuals who are student-centered, who research and question what has been learned, learn by doing and experiencing, and internalize and make sense of the information they have learned.

Although the studies showing the results of the teaching practice related to flipped learning in the literature are generally positive, they cannot provide definite data in terms of its effect on student success. In addition, there is a limited number of studies on nursing skills teaching related to the Flipped Learning method. In our country, there is no teaching example related to flipped learning in nursing education. However, the requirements and conditions include investigating the application and use of new models such as flipped learning; It was decided to carry out this research because it requires the collection of data on whether the application of this learning method is appropriate in nursing education at the universal and national level, especially in nursing skills training.

ELIGIBILITY:
Inclusion Criteria:

* Students who are in the 1st year of the Faculty of Nursing
* Students who will take the Nursing Fundamentals course
* Students who agreed to participate in the study

Exclusion Criteria:

* Nursing students who refused to participate in the study
* Health vocational high school graduate students
* Students who take the Nursing Fundamentals course from below

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Measuring Nursing Students' Academic Achievement Levels | To be measured at the end of the study (4 weeks later)
  Students in the control and study group will fill out the Student Introductory Information Form to explain the characteristics of the students.
  Afterwards, the Theoretical Information Evaluation Form, prepared in line with the aims and objectives of the course, will evaluate the theoretical information given to the students and will consist of multiple choice questions.
Measuring Nursing Students' Skill Levels | To be measured at the end of the study (4 weeks later)
  Arterial Blood Pressure Measurement, Pulse Counting, Respiratory Counting and Body Temperature Measurement Skill Checklists from the "Vital Signs" unit will be used to evaluate the skill levels of nursing students participating in the study. Validity and reliability studies will be conducted for each Skill Checklist to be used.

CONTACTS AND LOCATIONS:
Overall Officials: Nesrin OĞURLU, PhD Student, Study Chair — Aydın Adnan Menderes University Aydın Vocational School of Health Services; Gülengün TÜRK, Prof.Dr., Study Director — Aydın Adnan Menderes University Faculty of Nursing, Department of Nursing Fundamentals
Locations (1):
- Aydın Adnan Menderes University, Aydin, Efeler/ Aydın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Result] Choi J, Lee SE, Bae J, Kang S, Choi S, Tate JA, Yang YL. Undergraduate nursing students' experience of learning respiratory system assessment using flipped classroom: A mixed methods study. Nurse Educ Today. 2021 Mar;98:104664. doi: 10.1016/j.nedt.2020.104664. Epub 2020 Nov 11. PMID 33218906
- [Result] Gu M, Sok SR. Effects of Simulation Practicum Using Flipped Learning for Korean Nursing Students. Int J Environ Res Public Health. 2020 Sep 18;17(18):6829. doi: 10.3390/ijerph17186829. PMID 32962057
- [Result] Kim HS, Kim MY, Cho MK, Jang SJ. Effectiveness of applying flipped learning to clinical nursing practicums for nursing students in Korea: A randomized controlled trial. Int J Nurs Pract. 2017 Oct;23(5). doi: 10.1111/ijn.12574. Epub 2017 Jul 25. PMID 28741796
- [Result] Kim YM, Yoon YS, Hong HC, Min A. Effects of a patient safety course using a flipped classroom approach among undergraduate nursing students: A quasi-experimental study. Nurse Educ Today. 2019 Aug;79:180-187. doi: 10.1016/j.nedt.2019.05.033. Epub 2019 May 23. PMID 31153088
- [Result] Hampton D, Welsh D, Wiggins AT. Learning Preferences and Engagement Level of Generation Z Nursing Students. Nurse Educ. 2020 May/Jun;45(3):160-164. doi: 10.1097/NNE.0000000000000710. PMID 31219957